CLINICAL TRIAL: NCT00912119
Title: Pharmacokinetics of Epsilon-Aminocaproic Acid in Children Undergoing Craniofacial Reconstruction Surgery
Brief Title: Amicar Pharmacokinetics of Children Having Craniofacial Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paul Stricker (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other); Thomas B. and Jeannette E. Laws McCabe Fund Pilot Award (Unknown)
Responsible Party: Sponsor-Investigator, Paul Stricker, Assistant Professor for the University of Pennsylvania School of Medicine and The Children's Hospital of Philadelphia, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-007017
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Craniosynostosis
Keywords: craniofacial surgery; pharmacokinetics; cranial vault abnormalities; homologous blood products; wide scalp dissections; transfusion requirements
MeSH Terms: conditions — Craniosynostoses | interventions — Aminocaproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Group A - Low Dose
  Interventions: Drug: Epsilon-Aminocaproic Acid
- Group B (Experimental): Group B - Intermediate Dose
  Interventions: Drug: Epsilon-Aminocaproic Acid
- Group C (Experimental): Group C - High Dose
  Interventions: Drug: Epsilon-Aminocaproic Acid
- Group D (Experimental): Group D - Extra Low
  Interventions: Drug: Epsilon-Aminocaproic Acid

INTERVENTIONS:
Drug: Epsilon-Aminocaproic Acid — Group C (high dose) will receive a loading dose of EACA of 100 mg/kg over ten minutes followed by a continuous EACA infusion at 40 mg/kg/hr, which will be continued until the end of surgery.
  Other Names: Amicar; 6-aminohexanoic acid
  Arms: Group C
Drug: Epsilon-Aminocaproic Acid — Group A (low dose) will receive a loading dose of EACA of 25 mg/kg over ten minutes followed by a continuous EACA infusion at 10 mg/kg/hr, which will be continued until the end of surgery
  Other Names: Amicar; 6-aminohexanoic acid
  Arms: Group A
Drug: Epsilon-Aminocaproic Acid — Group B (intermediate dose) will receive a loading dose of EACA of 50 mg/kg over ten minutes followed by a continuous EACA infusion at 20 mg/kg/hr, which will be continued until the end of surgery
  Other Names: Amicar; 6-aminohexanoic acid
  Arms: Group B
Drug: Epsilon-Aminocaproic Acid — Group D (extra low dose) will receive a loading dose of EACA of 12.5 mg/kg over ten minutes followed by a continuous EACA infusion at 5 mg/kg/hr, which will be continued until the end of surgery
  Other Names: Amicar; 6-aminohexanoic acid
  Arms: Group D

SUMMARY:
Craniofacial reconstruction surgery involves a surgical approach to the craniofacial region to repair cranial vault and facial deformities. The surgery is extensive, often requiring wide scalp dissections and multiple osteotomies and has been associated with significant morbidity. Some of the most severe and commonly seen problems are associated with the rate and extent of blood loss.

Efforts to minimize surgical bleeding may translate to reduced transfusion requirements and a lessening of associated risks Epsilon-aminocaproic acid (EACA), an inhibitor of fibrinolysis, reduces transfusion requirements in children undergoing procedures on cardiopulmonary bypass (CPB), as well as in older children undergoing spinal surgery for scoliosis (1-6).

Before controlled studies to assess efficacy of EACA in a craniofacial surgical population can be done, appropriate pharmacokinetic (PK) data are needed to determine the optimal dosing strategy. PK data exist for EACA in children undergoing operations on CPB and hypothermia.

The aim of this study is to determine the pharmacokinetics of EACA in infants and children undergoing craniofacial reconstruction procedures.

DETAILED DESCRIPTION:
Craniosynostosis is the condition in which there is premature fusion of one or more of these sutures between the bones of the skull. Craniosynostosis limits the ability of the cranial vault to expand to accommodate the rapidly growing brain in infancy and early childhood. Deformation of skull shape results as cranial vault expansion occurs in areas of the skull that have not abnormally fused. Left uncorrected, craniosynostosis may adversely impact neurologic and psychosocial development. In some cases, increased intracranial pressure may also result.

Craniofacial (CF) reconstruction procedures to treat craniosynostosis are undertaken in young children to improve appearance, prevent functional disturbances, and enhance psychosocial development. Optimal surgical results are achieved when these procedures are performed in infancy. These procedures are extensive, often requiring wide scalp dissections and multiple osteotomies and have been associated with significant morbidity. Reported complications include massive blood loss, intraoperative cardiac arrest, transfusion reactions, venous air embolism, hypotension, coagulopathy, bradycardia, postoperative seizures, surgical site infections, facial swelling, and unplanned postoperative mechanical ventilation (7-13). Many of the most severe and commonly seen problems are associated with the rate and extent of blood loss.

Intraoperatively, the presence of hyperfibrinolysis has been demonstrated in children undergoing CF reconstruction procedures (8,14), although the extent of its contribution to bleeding is unclear.

Epsilon-aminocaproic acid (EACA), another inhibitor of fibrinolysis, is an attractive alternative. EACA is a synthetic lysine analog that blocks the lysine binding sites on plasminogen, resulting in antifibrinolytic activity through inhibition of plasmin formation.

We have chosen to study EACA in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of every race and ethnicity ages 2 months- 24 months
2. Diagnosis - Craniosynostosis (including syndromic craniosynostosis)
3. Surgical procedure - Pediatric patients undergoing craniofacial reconstruction procedures involving a craniotomy
4. Written informed parent/guardian consent

Exclusion Criteria:

1. Children with known or suspected hypersensitivity reaction to epsilon-aminocaproic acid
2. Subjects who do not have a parent or legal guardian who speaks English
3. Presence of a known coagulation abnormality
4. Presence of hematuria
5. Presence of a preoperative coagulation test abnormality (PT or PTT outside of normal range)
6. Known history of a coagulation disorder in either parent. Children in whom this history is not available (e.g., adopted children) will be eligible for study inclusion.
7. History of abnormal renal function
8. Serum creatinine or blood urea nitrogen (BUN) value outside of normal range (collected within 30 days of proposed EACA administration)
9. Initial intra-operative serum creatinine or BUN value outside of normal range
10. Children undergoing strip craniectomy for sagittal craniosynostosis
11. Presence of a preexisting neurologic deficit, seizure disorder, or other neurologic disorder
12. History of congenital cardiac disease (does not include patent ductus arteriosis, patent foramen ovale, or spontaneously closed muscular ventricular septal defect)
13. Children having other surgical procedures performed in addition to craniofacial reconstruction surgery
14. Preoperative laboratory abnormalities that indicate clinically significant hematologic disease (collected within 30 days of proposed EACA administration):

    Hemoglobin < 9 gm/dL Platelet count < 100,000/mm3
15. Any investigational drug use within 30 days prior to proposed EACA administration.
16. Wards are not eligible for study
17. Children who have been previously enrolled in this study may not be enrolled again.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters of EACA including clearance, AUC0-∞, half-life, and volume of distribution | 80 hours

SECONDARY OUTCOMES:
Volume of homologous blood (mL/kg) transfused postoperatively | 72 hours
Volume of homologous blood (mL/kg) transfused intraoperatively | 6 hours
Safety and tolerability of EACA based on the occurrence of Adverse Events | 720 hours
Potentially defining a Maximum Tolerated Dose (MTD) for EACA in the stated population | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stricker, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States